CLINICAL TRIAL: NCT00393380
Title: A Phase II Study of Parathyroid Hormone Following Myeloablative Sequential Unrelated Cord Blood Transplantation
Brief Title: Study of Parathyroid Hormone Following Sequential Cord Blood Transplantation From an Unrelated Donor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped because of toxicity concerns.
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 435; U54HL081030-02 (NIH); NCT00579722 (obsolete NCT alias)
Record Dates: First submitted 2006-10-25; First posted 2006-10-27 (Estimated); Results first posted 2012-12-07 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia, Myeloid, Chronic; Anemia, Aplastic; Myelofibrosis; Lymphoma; Hodgkin Disease; Leukemia, Lymphocytic, Chronic; Leukemia, Myelocytic, Acute; Leukemia, Lymphocytic, Acute
Keywords: Myelogenous Leukemia, Chronic; Myelodysplasia; Parathyroid Hormone; Umbilical Cord Blood Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Anemia, Aplastic; Primary Myelofibrosis; Lymphoma; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts | interventions — Parathyroid Hormone; Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Parathyroid Hormone (teriparatide) (Experimental): Parathyroid hormone after double umbilical cord blood transplant.
  Interventions: Drug: Parathyroid Hormone (teriparatide)

INTERVENTIONS:
Drug: Parathyroid Hormone (teriparatide) — Day +1: PTH 40 mcg, Day +2: PTH 60 mcg, Day +3: PTH 80 mcg, Day +4 to Day +29 or until ANC>2000/microL: PTH 100 mcg
  Other Names: Parathyroid hormone; PTH; teriparatide

SUMMARY:
The purpose of this study is to determine whether the addition of parathyroid hormone after a sequential cord blood transplant will improve engraftment, which is the ability of the transplanted stem cells to grow and to successfully begin producing new blood cells.

DETAILED DESCRIPTION:
In this phase II, single stage study, participants will include 40 adults who are candidates for a hematopoietic stem cell transplant. All participants will undergo a sequential cord blood transplant using a well-known myeloablative regimen of fludarabine, cyclophosphamide, and total body irradiation, which is appropriate for those individuals who are likely to benefit from an ablative regimen. Tacrolimus will be combined with mycophenolate mofetil (MMF) for the graft-versus-host disease (GVHD) prophylaxis regimen. Parathyroid hormone (PTH) will be added to this regimen in an attempt to improve engraftment. PTH is an approved drug with minimal side effects in individuals with osteoporosis; the dose of PTH has been determined from a phase I study in individuals with hematologic cancer.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses:

  1. Chronic myelogenous leukemia (CML) accelerated phase or second stable phase; individuals in the first chronic phase are eligible if they have resistance to imatinib
  2. Myelodysplasia
  3. Aplastic anemia that is not responding to immunosuppressive therapy
  4. Myelofibrosis, either primary or secondary to polycythemia vera
  5. Relapsed lymphoma or Hodgkin's disease
  6. Stage III/IV chronic lymphocytic leukemia (CLL), relapsed after or refractory to at least one fludarabine containing regimen
  7. Acute myelogenous leukemia (AML) or acute lymphoblastic leukemia (ALL) in complete remission (CR) 2 or greater, or CR 1 with high risk features
* No prior autologous stem cell transplant
* Eastern Cooperative Oncology Group (ECOG) performance status of less than 2
* Lack of 6/6 or 5/6 matched related donor OR lack of 10/10 matched unrelated donor OR no available donor in the appropriate time frame to perform a potentially curative stem cell transplant
* Diffusing capacity of the lung for carbon monoxide (DLCO) greater than 50% of predicted value
* Left ventricular ejection fraction (LVEF) greater than 50% of predicted value
* Calcium levels less than 10.5 mg/dl
* Phosphate levels greater than 1.6 mg/dl

Exclusion Criteria:

* Heart disease, as determined by symptomatic congestive heart failure, radionuclide ventriculogram (RVG), or echocardiogram-determined LVEF of less than 50%, active angina pectoris, or uncontrolled high blood pressure
* Pulmonary disease, as determined by severe chronic obstructive lung disease, symptomatic restrictive lung disease, or corrected DLCO of less than 50% of predicted value
* Kidney disease, as determined by serum creatinine levels greater than 2.0 mg/dl
* Liver disease, as determined by serum bilirubin levels greater than 2.0 mg/dl (except in the case of Gilbert's syndrome or hemolytic anemia in which the bilirubin can be elevated greater than 2.0mg/dl), SGOT or SGPT greater than 3 times the upper limit of normal
* Neurologic disease, as determined by symptomatic leukoencephalopathy, active central nervous system (CNS) cancer, or other neuropsychiatric abnormalities that may prevent transplantation (previous CNS cancer and presently in CR is acceptable)
* HIV antibodies
* Uncontrolled infection
* Pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2006-09; Primary Completion 2009-11 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen K. Ballen, MD, Principal Investigator — Massachusetts General Hospital; Joseph Antin, MD, Principal Investigator — Dana-Farber Cancer Institute; David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Elizabeth J Shpall, MD, Principal Investigator — MD Anderson Cancer Research Center; Colleen Delaney, MD, Principal Investigator — Fred Hutchinson Cancer Center; Ram Kamble, MD, Principal Investigator — Baylor College of Medicine; Katarzyna Jamieson, M.D., Principal Investigator — University of Florida; Philip McCarthy, M.D., Principal Investigator — Roswell Park Cancer Institute; Edward Ball, M.D., Principal Investigator — University of California, San Diego; Richard Maziarz, M.D., Principal Investigator — Oregon Health and Science University
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Ballen K, Mendizabal AM, Cutler C, Politikos I, Jamieson K, Shpall EJ, Dey BR, Attar E, McAfee S, Delaney C, McCarthy P, Ball ED, Kamble R, Avigan D, Maziarz RT, Ho VT, Koreth J, Alyea E, Soiffer R, Wingard JR, Boussiotis V, Spitzer TR, Antin JH. Phase II trial of parathyroid hormone after double umbilical cord blood transplantation. Biol Blood Marrow Transplant. 2012 Dec;18(12):1851-8. doi: 10.1016/j.bbmt.2012.06.016. Epub 2012 Jul 2. PMID 22766223

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen patients were enrolled on the study between October 25, 2006 and March 27, 2008 from three centers. Dana Farber Cancer Institute enrolled 10 patients, University of Florida enrolled 2 patients and Massachusetts General Hospital enrolled 1 patient.
Pre-assignment Details: Thirteen patients who were enrolled proceeded to the cord blood transplant.
Period: Overall Study
Arm/Group | Parathyroid Hormone (Teriparatide)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Parathyroid Hormone (Teriparatide)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 2
Age Continuous [Median (Full Range); unit: years] — Median Age at Transplant
  years | 39 [25 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race among patients transplanted.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 10
    More than one race | 2
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Neutrophil Engraftment (Defined as an Absolute Neutrophil Count [ANC] Greater Than 500)
Description: Median time to neutrophil engraftment (defined as an absolute neutrophil count [ANC] greater than 500)
Time Frame: Statistic is calculated at Day 42 but ANC counts are measured daily up through discharge.
Population: 13 patients received the transplant.
Measure: Median (Full Range); unit: days
Arm/Group | Parathyroid Hormone (Teriparatide)
Number analyzed (Participants) | 13
days | 30 [19 to 37]

2. Secondary Outcome: Cumulative Incidence of Acute GVHD Grades II-IV at Day 100
Description: Cumulative Incidence of Acute GVHD Grades II-IV at day 100
Time Frame: Measured at Day 100
Population: 13 patients were transplanted
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parathyroid Hormone (Teriparatide)
Number analyzed (Participants) | 13
percentage of participants | 38.5 [10.3 to 66.7]

3. Secondary Outcome: Cumulative Incidence of Chronic GVHD
Description: Cumulative Incidence of Chronic GVHD
Time Frame: Measured at 2 years
Population: 13 patients were transplanted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parathyroid Hormone (Teriparatide)
Number analyzed (Participants) | 13
percentage of participants | 38.5 [8.1 to 68.9]

4. Secondary Outcome: Platelet Engraftment (Greater Than 20,000)
Description: Platelet engraftment (greater than 20,000)
Time Frame: Measured at Day 180
Population: 13 patients were transplanted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parathyroid Hormone (Teriparatide)
Number analyzed (Participants) | 13
percentage of participants | 46.2 [17.0 to 76.0]

5. Secondary Outcome: 100-day Transplant-related Mortality
Description: 100-day transplant-related mortality
Time Frame: Measured at Day 100
Population: 13 patients were transplanted
Measure: Number; unit: participants
Arm/Group | Parathyroid Hormone (Teriparatide)
Number analyzed (Participants) | 13
participants | 4

6. Secondary Outcome: Cumulative Incidence of Relapse
Description: Cumulative Incidence of Relapse
Time Frame: Measured at 2 years
Population: 13 patients were transplanted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parathyroid Hormone (Teriparatide)
Number analyzed (Participants) | 13
percentage of participants | 15.4 [0.0 to 36.2]

7. Secondary Outcome: Overall Survival
Description: Overall Survival
Time Frame: Measured at 2 years
Population: 13 patients were transplanted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parathyroid Hormone (Teriparatide)
Number analyzed (Participants) | 13
percentage of participants | 38.5 [14.1 to 62.8]

8. Secondary Outcome: Disease-free Survival
Description: Disease-free survival
Time Frame: Measured at 1 year
Population: 13 patients were transplanted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Parathyroid Hormone (Teriparatide)
Number analyzed (Participants) | 13
percentage of participants | 38.5 [14.1 to 62.8]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Parathyroid Hormone (Teriparatide)
Serious Adverse Events (participants affected / at risk) | 8/13
Other Adverse Events (participants affected / at risk) | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parathyroid Hormone (Teriparatide) (N=13)
Death (General disorders) | 8 (8) — Death
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parathyroid Hormone (Teriparatide) (N=13)
Death (General disorders) | 8 (8)

LIMITATIONS AND CAVEATS:
The study was closed prematurely due to early mortality and lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No